CLINICAL TRIAL: NCT02681952
Title: A Multicenter, Randomized, Open-labeled, Cross-over, Active-controlled, Phase IV Clinical Trial to Evaluate the Preference of Formulation and the Efficacy and Safety of Renamezin and Kremezin in Pre-dialysis Patients With Chronic Renal Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DW_RNMZ_401
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

ARMS (2):
- Renamezin->Kremezin (Active Comparator)
  Interventions: Drug: Renamezin capsule; Drug: Kremezin granule
- Kremezin->Renamezin (Active Comparator)
  Interventions: Drug: Renamezin capsule; Drug: Kremezin granule

INTERVENTIONS:
Drug: Renamezin capsule
Drug: Kremezin granule

SUMMARY:
A Multicenter, Randomized, Open-labeled, Cross-over, Active-controlled, Phase IV Clinical Trial to Evaluate the Preference of Formulation and the Efficacy and Safety of Renamezin and Kremezin in Pre-dialysis Patients With Chronic Renal Failure

ELIGIBILITY:
Inclusion Criteria:

* pre-dialysis patients with chronic renal failure stage
* patient for holding the stable state in serum creatinine 2.0mg/dl - 5.0mg/dl of MDRD GFR 15-60ml/min/1.73m2 for 3 months before screening
* patients haven't experienced dose spherical carbon adsorbent for 3months before screening
* patients who were no noticeable change for 4weeks before screening and are expected to change is not needed during therapy in the therapy of chronic renal failure(type of blood pressure medication and dose -related, diet therapy)
* patients spontaneously written consent to participate in this clinical trial

Exclusion Criteria:

* patients with passes through the digestive tract disorders
* patients with uncontrolled constipation symptoms
* kidney transplant patients
* patients who are taking immunosuppressive drugs
* patients suffering from digestive tract ulcers and esophageal varices
* patients with uncontrolled hypertension
* patients hospitalized with cardiovascular disease within 3 months of the screening
* patients with current infections
* patients who do not fulfill therapies of chronic renal failure (taking medicine and diet) as appropriate
* patients with hepatic impairment (2.5 times greater than the upper limit of normal levels of AST, ALT)
* uncontrolled diabetes (HbA1c > 10 % or a fasting glucose > 180mg / dL)
* patients with malignant tumors (However, if you do not relapse within five years after completion of therapy can be registered)
* pregnant women, nursing mothers
* those who do not agree to a contraceptive method allowed for the possibility of pregnancy in women
* patients participating in another clinical trial in addition to the current clinical trial
* subjects with dependency on drugs or alcohol
* subjects who took any other investigational drugs within 30 days before participating this clinical trial study
* patients expected to starting the dialysis within three months
* other patients deemed unsuitable tester

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Preference of formulation | 24weeks
  questionnaire

SECONDARY OUTCOMES:
Serum Creatinine | 12weeks, 24weeks
Serum Indoxyl sulfate | 12weeks, 24weeks
Cystatin-C | 12weeks, 24weeks
estimated GFR(Glomerular Filtration Rate) | 12weeks, 24weeks
  MDRD GFR

CONTACTS AND LOCATIONS:
Overall Officials: Bumseok Kim, Professor, Principal Investigator — Sevrance Hospital of Yonsei University
Locations (1):
- Sevrance Hospital of Yonsei University, Seoul, Seodaemun, South Korea

REFERENCES:
- [Derived] Kee YK, Han SY, Kang DH, Noh JW, Jeong KH, Kim GH, Kim YW, Kim BS. Comparison of Different Types of Oral Adsorbent Therapy in Patients with Chronic Kidney Disease: A Multicenter, Randomized, Phase IV Clinical Trial. Yonsei Med J. 2021 Jan;62(1):41-49. doi: 10.3349/ymj.2021.62.1.41. PMID 33381933